CLINICAL TRIAL: NCT04590482
Title: Use of Letrozole Pretreatment With Misoprostol for Induction of Abortion in First Trimester Missed Abortion
Brief Title: Letrozole Pretreatment With Misoprostol Induction of Abortion in First Trimester Missed Abortion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shereen Rady Abou El-fetouh (Other)
Responsible Party: Sponsor-Investigator, Shereen Rady Abou El-fetouh, principal investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Letrozole /pretreatment
Record Dates: First submitted 2020-08-23; First posted 2020-10-19 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Missed Abortion
MeSH Terms: conditions — Abortion, Missed | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: participant- care provider -investigator- outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- letrozole then misoprostol (Experimental): description:letrozole 2.5 mg each 12hours for 2 days at home followed by misoprostol 800mcg vaginally at hospital repeated after 4 hours if needed
  Interventions: Drug: letrozole
- placebo then misoprostol (Placebo Comparator): Description:placebo each 12 hours for 2days at home followed by 800mcg misoprostol vaginally at hospital and repeat dose after 4 hours if needed
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: letrozole — Letrozole 2.5 mg each 12 hours for 2 days followed by vaginal misoprostol 800 mcg for induction of abortion
  Arms: letrozole then misoprostol
Drug: placebo — placebo given twice daily for 2 days followed by 800mcg misoprostol vaginally to induce abortion
  Arms: placebo then misoprostol

SUMMARY:
this study will compare the efficacy of using letrozole pre treatment before misoprostol versus using misoprostol only in the induction of first trimester missed abortion.

DETAILED DESCRIPTION:
Intervention type: drug

Intervention name: letrozole then misoprostol

Description :letrozole 2.5mg twice per day for 2days then misoprostol 800mcg for all patients to induce abortion

Arm group label:study group

Intervention type :drug

Intervention name:placebo then misoprostol

Description : placebo for 2days then 800mcg misoprostol to all patients to induce abortion

Arm group label: control group

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age more than 18 years old.
2. Gestational age less than 13 weeks confirmed by ultrasound scan on day 1 of the study.
3. Hemoglobin >10 g/dl
4. Missed abortion

Exclusion Criteria:

1. Mullerian Uterine anomalies as septate, bicornuate uterus.
2. Fibroid uterus.
3. Coagulopathy.
4. Medical disorder that contraindicate induction of abortion.
5. Allergy to misoprostol or letrozole.

   -

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Ages of eligibility :18years and older
  sex eligibility :female
Enrollment: 110 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-03-16 (Estimated); Study Completion 2021-05-08 (Estimated)

PRIMARY OUTCOMES:
Complete abortion | 6 hours
  incidence of complete abortion without the need of surgical evacuation among 110patients in which 55 of patients took letrozole before misoprostol and the other 55 patients took placebo before misoprostol

SECONDARY OUTCOMES:
surgical evacuation | 6 hours
  surgical evacuation for the remnants of conception among 110 patients in which 55 took letrozole before misoprostol and other 55 patients who took placebo before misoprostol

CONTACTS AND LOCATIONS:
Overall Officials: shereen khedr, Principal Investigator — AinShams University

IPD SHARING:
Plan to Share IPD: No